CLINICAL TRIAL: NCT02038855
Title: International Latino Research Partnership
Acronym: ILRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hospital Vall d'Hebron (Other); Universidad Autonoma de Madrid (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHA-IRB-0910/06/12; R01DA034952-01A1 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-01-17 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Substance Use (Drugs, Alcohol)
Keywords: Dual-diagnosis; Latino; Mental health; Substance use; HIV risk
MeSH Terms: conditions — Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IIDEA (Active Comparator): Patients in the Integrated Intervention for Dual Problems and Early Action (IIDEA) arm will receive the 10 session intervention administered in person and via telephone.
  Interventions: Behavioral: Integrated Intervention for Dual Problems and Early Action
- Usual Care (No Intervention): Patients in this arm receive usual care for dual-diagnosis symptoms of mental health and substance use. They receive 5 check-in calls from a care manager to assess safety.

INTERVENTIONS:
Behavioral: Integrated Intervention for Dual Problems and Early Action — Integrated Intervention for Dual Problems and Early Action (IIDEA) includes psycho-education, Cognitive Behavioral Therapy and mindfulness; identifies triggers and challenging thoughts; provides motivational techniques for reducing substance use and/or smoking cravings; incorporates cognitive restructuring to identify and correct negative thinking patterns influenced by depression, anxiety and/or trauma; and includes self-monitoring of thoughts and risk behaviors that contribute to substance use, smoking and increased HIV risk.
  Arms: IIDEA

SUMMARY:
Through a grant funded by the National Institute on Drug Abuse (NIDA) the Center for Multicultural Mental Health Research at Cambridge Health Alliance is testing a screening and intervention project designed to improve the quality of care for Latino patients with comorbid mental health and substance use problems. We will first test a screening of comorbid problems with patients identified in mental health as well as primary health care. Building on that work, we will test the feasibility, acceptability and efficacy of the "Integrated Intervention for Dual Problems and Early Action" (IIDEA) intervention addressing mental health, substance use, and prevention of HIV, as well as a smoking cessation supplement. The project is being conducted in Massachusetts as well as at two sites in Spain. As such, the proposed ILRP multi-site international project is a critical step towards developing models of integrated care for the large and diverse Latino migrant population and more broadly towards understanding how best to integrate evidence-based assessment and treatments for co-occurring substance and mental health problems and HIV risks.

DETAILED DESCRIPTION:
Our study aims to conduct behavioral health services research focused on rapid screening and referral; as well as testing the feasibility, acceptability and efficacy of integrated behavioral health services in primary care clinics for migrant Latinos with co-occurring substance use and mental health problems, and increased risk of HIV.

A key activity for the first phase, the screening project, is administering a screener to at least 450 Latino migrant patients across the 3 sites (n=150 each in Boston, Madrid, and Barcelona) from primary care and behavioral health (substance abuse and mental health) services. We intend to test the referral process for screened participants in need of treatment to identify barriers and streamline the process. We will analyze data to optimize the screening battery and protocol to use in Phase 2, the IIDEA intervention.

In Phase 2, we intend to enroll, randomize and collect data on 360 total patients across the 3 sites - 180 in the intervention condition and 180 in the control condition (120 in each site, 60 in the intervention condition and 60 in the control condition). The 10 session IIDEA intervention will be offered to Latino patients by trained clinicians with at least a Masters level of training. The intervention is designed to help patients to address and prevent mental health and substance use problems and will be culturally adapted to Latino populations in Boston, Madrid and Barcelona. Usual care - the control group - receives treatment as usual, for patients in primary care identified with a mental health or substance use problem. 5 Research interviews will be conducted to assess outcomes, for patients in both the intervention and usual care arms.

ELIGIBILITY:
Inclusion Criteria:

* Latino migrants
* Must speak English or Spanish
* 18-70 years of age
* Screen positive to at least one substance use and one mental health problem

Exclusion Criteria:

* Current or recent (last 3 months) substance use treatment (more than 1 visit with a provider at a behavioral health clinic)
* Planning to receive behavioral health services (i.e., have an appointment scheduled in the next 2 months)
* Evidence that the patient lacks capacity to consent to the study
* Evidence of current suicidal risk or harm to others (affirmative responses to questions 4 and/or 5 on Paykel suicide questionnaire)- patient can be rescreened in 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI) - Alcohol (change) | Baseline, 2 months, 4 months, 6 months, 12 months
  The ASI is a semi-structured interview designed to address seven potential problem areas in substance-abusing patients; this outcome measure refers to the Alcohol problem area.
Addiction Severity Index (ASI) - Drugs (change) | Baseline, 2 months, 4 months, 6 months, 12 months
  The ASI is a semi-structured interview designed to address seven potential problem areas in substance-abusing patients; this outcome measure refers to the Drug problem area.
Change on Urine Drug Test (change) | Baseline, 2 months, 4 months, 6 months, 12 months
  Technical analysis of a biological specimen (urine) to determine the presence or absence of specified parent drugs or their metabolites.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder 7-item (GAD-7) Scale (change) | Baseline, 2 months, 4 months, 6 months, 12 months
  The GAD-7 is a questionnaire for screening and severity measuring of generalized anxiety disorder (GAD).
PTSD Checklist for DSM-V (PCL-5) | Baseline, 2 months, 4 months, 6 months, 12 months
  The PCL-5 is is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD.
Patient Health Questionnaire (PHQ-9) (change) | Baseline, 2 months, 4 months, 6 months, 12 months
  The PHQ-9 is a 9-item screening questionnaire to determine level of depressive disorder.
Hopkins Symptom Checklist-20 | Baseline, 2 months, 4 months, 6 months, 12 months
  The HSCL-20 is a symptom inventory for depression that indicates severity of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Alegria, Ph.D., Principal Investigator — CMMHR, Cambridge Health Alliance and Harvard Medical School; Enrique Baca-Garcia, Ph.D., Principal Investigator — Universidad Autonoma de Madrid; Francisco Collazos, MD, Principal Investigator — Vall d'Hebron University Hospital
Locations (3):
- Cambridge Health Alliance, Somerville, Massachusetts, United States
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona, Catalonia
  - Universidad Autonoma de Madrid Medical School, Madrid

REFERENCES:
- [Derived] Levison JH, Alegria M, Wang Y, Markle SL, Fuentes L, Mejia DL, Tarbox A, Albarracin Garcia L, Cellerino L, El-Bassel N. High HIV/STI Test Acceptance Through a Behavioral Health Encounter in Latino Immigrants with Substance Use and Mental Health Problems. AIDS Behav. 2019 Apr;23(4):835-846. doi: 10.1007/s10461-019-02413-y. PMID 30737609
- [Derived] Alegria M, Falgas-Bague I, Collazos F, Carmona Camacho R, Lapatin Markle S, Wang Y, Baca-Garcia E, Le Cook B, Chavez LM, Fortuna L, Herrera L, Qureshi A, Ramos Z, Gonzalez C, Aroca P, Albarracin Garcia L, Cellerino L, Villar A, Ali N, Mueser KT, Shrout PE. Evaluation of the Integrated Intervention for Dual Problems and Early Action Among Latino Immigrants With Co-occurring Mental Health and Substance Misuse Symptoms: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jan 4;2(1):e186927. doi: 10.1001/jamanetworkopen.2018.6927. PMID 30646205
- See also: Project Website — http://www.multiculturalmentalhealth.org/International_Latino_Research_Partnership.asp